CLINICAL TRIAL: NCT00547404
Title: An Open Label, Multicenter Phase I Study To Evaluate Safety and Efficacy of P276-00 in Subjects With Relapsed and Relapsed/Refractory Multiple Myeloma
Brief Title: Phase I Study for Safety and Efficacy of P276-00 in Subjects With Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not to expose the patients to subtherapeutic dose
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Dr Himanshu Parikh, Piramal Life Sciences Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/11/07
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: P276-00 — IV drug infusion over a period of 30 min on day 1,4,8 and 11 in21 day cycle for 6 cycles

SUMMARY:
This research study is a Phase I/II clinical trial. It is done to determine the best doses that the investigational drug (P276-00) can be used safely. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more information about it such as; the safest dose to use, the side effects it may cause and if it is effective for treating relapsed/refractory multiple myeloma.

A majority of multiple myeloma patients overexpress a protein that plays a role in regulating the body's cell cycle called Cyclin D1. The study drug P276-00 is a Cyclin D1 inhibitor under investigation in the treatment of solid tumors. The researchers therefore believe that Cyclin D1 should be studied as a therapeutic target in myeloma. In this research study, we are looking for the highest dose of P276-00 that can be given safely and to see how well it works

DETAILED DESCRIPTION:
The pre clinical data demonstrated that P276-00 is a selective Cdk4-D1 and Cdk1-B inhibitor with potent cytotoxic effects against MM cells including sensitive (MM1.S, RPMI 8226, OPM1, OPM2) and resistant (MM1.R, Dox-40, LR5) to conventional chemotherapy as well as in mouse xenograft models. The IC50 for this effect is between 300-1000 nM in vitro, and potential doses to be evaluated in the clinical study can achieve these concentrations. This evidence supports a rationale for evaluating the effects of P276-000 in patients with relapsed/refractory MM in order to determine safety and tolerability as well as pharmacokinetics and potential efficacy. The current study design allows for adequate assessment of patient safety in terms of the potential adverse effects of P276-00.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject previously diagnosed with multiple myeloma based either on the standard or the International Myeloma Foundation (IMF) diagnostic criteria as defined in Appendix A 2. Subjects must have relapsed or relapsed/refractory disease after at least 2 prior lines of therapy as defined in Appendix D 3. Monoclonal protein in the serum of ³ 1 gm/dL or monoclonal light chain in the urine protein electrophoresis of ³ 200 mg/ 24 hours, or measurable light chains by free light chain assay of ³ 10 mg/dL, or measurable plasmacytoma 4. Age ≥ 18 years at the time of signing the informed consent form 5. ECOG performance status < 2 6. Life expectancy > 3 months 7. Subjects must have the following laboratory parameters:

  * Hemoglobin > 8.0 gm/dL
  * Absolute neutrophil count (ANC) ≥1000 cells/mm3
  * Platelets count ≥ 50,000/mm3
  * Serum SGOT/AST <3.0 x institutional upper limits of normal (ULN)
  * Serum SGPT/ALT <3.0 x institutional upper limits of normal (ULN)
  * Serum creatinine <2.5mg/dL
  * Serum total bilirubin <1.5 x institutional upper limits of normal (ULN) 8. Woman of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months) with a negative serum pregnancy test. In addition, all sexually active woman of childbearing potential and men agreeing to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilised 9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* 1. Subjects having received radiotherapy, immunotherapy, chemotherapy and or biological agents like G-CSF in the 2 weeks prior to day 1 of study drug administration and have not recovered completely from the side effects of the earlier investigational agent 2. Subjects having received any other investigational agents within 2 weeks prior to the date of enrolment 3. History of allergic reactions attributed to compounds of similar chemical composition to P276-00 4. Subjects with a history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months 5. Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the subject has been disease-free for at least 3 years 6. Subjects with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, known cardiac ejection fraction <40%, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements 7. Women who are pregnant or nursing 8. Subjects known to be seropositive for the human immunodeficiency virus 9. Subjects requiring the use of concomitant medications that prolong the QT/QTc interval and/or are known to cause Torsades de Pointes (TdP) 10. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) in subjects with relapsed and relapsed/refractory Multiple Myeloma (MM) | 1year

SECONDARY OUTCOMES:
clinical response of P276-00 in subjects with relapsed and relapsed/refractory MM 2. Exploratory pharmacogenomic analysis of serum and molecular markers associated with P276-00 use in the study population | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Dana-Farber Cancer Institute; Sagar Lonial, MD, Principal Investigator — Winship Cancer Institute,Emory University; Sundar Jagannath, MD, Principal Investigator — St. Vincent's Comprehensive Cancer Center